CLINICAL TRIAL: NCT06075355
Title: Sagittal : Can Minimally Invasive Decompression Surgery Restore Sagittal Balance in a Patient Population With Sagittal Imbalance and Lumbar Spinal Stenosis
Brief Title: Can Minimally Invasive Decompression Surgery Restore Sagittal Balance in a Patient Population With Sagittal Imbalance and Lumbar Spinal Stenosis
Status: Not yet recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Sagittal
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lumbar Spinal Stenosis
Keywords: lumbar stenosis; sagittal imbalance; minimally invasive decompression surgery
MeSH Terms: conditions — Spinal Stenosis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
From adulthood onwards, the aging process manifests itself in the spine through loss of disc height and kyphotic deformity. As the general population ages, the prevalence of lumbar degenerative diseases and sagittal imbalance increases. Sagittal balance is a physiological alignment resulting from the effective muscular and ligamentary forces that place patients' heads harmoniously in line with their pelvis. Roussouly first classified this alignment by differentiating four types of balance in an asymptomatic population. He established a link between the varieties of sagittal balance of the spine, the sacral slope and the position of the pelvis in space. He went on to explain sagittal imbalance in the aging population suffering from degenerative diseases.

One of the most common lumbar degenerative diseases is lumbar spinal canal stenosis. Stenosis of the lumbar spinal canal is frequently associated with sagittal imbalance of the spine. Lumbar canal stenosis causes lumbar pain, leg pain, neurogenic intermittent claudication and bladder and rectal disorders. The severity of clinical symptoms increases linearly with progressive sagittal imbalance [8]. We represent the sagittal imbalance of the spine by a positive sagittal vertical axis (SVA) presented by patients to reduce the pressure exerted by the yellow ligament, which is hypertrophied in degenerative disease . Many have shown that this forward-flexing posture can be improved by simple decompression, and that this deformity corresponds to an analgesic position and not to a structural deformity. Little is known about the factors that influence alignment after lumbar canal decompression and short segment fusion.

This study therefore aims to elucidate some of the clinical and radiological factors likely to affect postoperative sagittal balance in patients undergoing simple minimally invasive decompression surgery and short segment fusion (1 or 2 levels).

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* French-speaking patients
* Patients undergoing minimally invasive lumbar decompression with or without one- or two-level arthrodesis
* Patients with preoperative sagittal imbalance measured on EOS images (sagittal vertebral axis > 50 mm)

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his or her data for this study
* Revision surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient suffering from lumbar stenosis, adressed for minimally invasive lumbar decompression between january, 1st 2014 and january 31st, 2020
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of sagittal balance after minimally invasive decompression surgery | 3 months
  Sagittal Vertebral axis mesurement before and after surgery

SECONDARY OUTCOMES:
barrey Ratio | 3 months
  mesurement of the Barrey Ratio before and after surgery
lumbar lordosis | 3 months
  mesurement of the lumbar lordosis before and after surgery
pelvic incidence | 3 months
  mesurement of the pelvic incidence before and after surgery
pelvic version | 3 months
  mesurement of the pelvic version before and after surgery
sacred gradient | 3 months
  mesurement of the sacred version before and after surgery
thoracic kyphosis | 3 months
  mesurement of the thoracic kyphosis before and after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Paris Saint Joseph, Paris, France